CLINICAL TRIAL: NCT02423330
Title: A Prospective Evaluation of the Strattice-LIFT to Treat Anal Fistula
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study terminated by sponsor
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14072904
Record Dates: First submitted 2015-04-17; First posted 2015-04-22 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Anal Fistula; Rectal Fistula; Fistula in Ano; Transsphincteric Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Strattice-LIFT (Experimental)
  Interventions: Device: Strattice-LIFT

INTERVENTIONS:
Device: Strattice-LIFT — Patients undergoing surgery for transsphincteric anal fistulas will undergo the Strattice-LIFT procedure. A standard LIFT procedure will be performed with the addition of Strattice placed into the intersphincteric space.

SUMMARY:
This clinical trial will evaluate the safety and efficacy of the Strattice-LIFT procedure to treat anal fistulas.

DETAILED DESCRIPTION:
The treatment of anal fistulas remains a challenging clinical problem. Fistulotomy is highly effective, but carries a significant risk of postoperative incontinence. A variety of surgical procedures that do not divide the sphincter muscle may be offered to patients, however none of them are as effective as fistulotomy.

The LIFT (ligation of intersphincteric fistula tract) procedure is a newer option for the treatment of transsphincteric fistulas. Initial results have been promising. However, some fistulas recur after the LIFT procedure because the divided ends of the fistula tract recanalize. Insertion of a barrier into the intersphincteric space may prevent this process. Strattice is acellular porcine dermis, will be used for this purpose.

This prospective trial will evaluate the safety and efficacy of the Strattice-LIFT procedure for the treatment of transsphincteric anal fistulas.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 22 years of age or older
2. Subject is willing to comply with study related procedures
3. Subject is not pregnant
4. Subject has a transsphincteric fistula
5. Subject is medically fit to undergo LIFT
6. Subject has a draining seton for a minimum of 6 weeks

Exclusion Criteria:

1. Crohn's disease
2. Pelvic radiation treatment
3. Known or suspected HIV/AIDS
4. Known sensitivity to pork products
5. Abscess or fistula etiology other than cryptoglandular
6. Abdominal malignancies
7. Patients with <1 year life expectancy
8. History of smoking
9. Known anorectal dysfunction (fecal incontinence)
10. Chronic use of steroids or other agents which may affect wound healing
11. ASA ≥ 2
12. Unable to consent to study
13. Unable to complete 1 year follow up

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Healing of the anal fistula | 6 months
  Healing is defined as the combination of patient reported lack of drainage and surgeon reported closure of the external opening

SECONDARY OUTCOMES:
Healing of the anal fistula | 1 year
  Healing is defined as the combination of patient reported lack of drainage and surgeon reported closure of the external opening
Postoperative Pain | 1 year
  Postoperative pain will be assessed at each postoperative visit with a visual analog scale
Complications | 1 year
  Postoperative complications such as infection/abscess, bleeding, urinary retention, new fistula, constipation, or fecal incontinence

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States